CLINICAL TRIAL: NCT04155450
Title: Effects of Extension Biased External Limb Loading in Addition to McKenzie Extension Protocol in Lumbar Derangement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2019/2
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Sciatica; Low Back Pain; Low Back Pain, Mechanical
Keywords: exercise; manipulation, spinal; rehabilitation; therapy, manual; manual therapy
MeSH Terms: conditions — Sciatica; Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant is unaware of the treatment group he is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie Extension with External Limb Loading Protocol (Experimental): Moist Heat Pack for 10 mins
  McKenzie Extension Exercise Protocol
  Static:
  1. Lying Prone
  2. Lying prone in extension
  3. Sustained extension
  4. Posture correction
     Dynamic:
  5. Extension in lying
  6. Extension in lying with clinician overpressure
  7. Extension mobilization
  8. Extension in standing
  Limb loading for basic stabilization progression of the lumbar extensors. Begin in the quadruped position and progress the intensity by
  1. Flexing one upper extremity
  2. Extending one lower extremity with a leg slide
  3. Extending one lower extremity by lifting it off the mat
  4. Flexing one upper extremity while extending contralateral lower extremity and then alternate to opposite extremities.
     Progress to prone position:
  5. Extending one lower extremity
  6. Extending both lower extremity
  Interventions: Other: Extension Biased External Limb Loading Exercises; Other: McKenzie Extension Exercise Protocol; Other: Moist Heat
- McKenzie Extension Group (Active Comparator): Moist Heat Pack for 10 mins
  McKenzie Extension Protocol Sequence
  Static:
  1. Lying Prone
  2. Lying prone in extension
  3. Sustained extension
  4. Posture correction
     Dynamic:
  5. Extension in lying
  6. Extension in lying with clinician overpressure
  7. Extension mobilization
  8. Extension in standing
  Interventions: Other: McKenzie Extension Exercise Protocol; Other: Moist Heat

INTERVENTIONS:
Other: Extension Biased External Limb Loading Exercises — Begin in the quadruped position and progress the intensity by
  1. Flexing one upper extremity
  2. Extending one lower extremity with a leg slide
  3. Extending one lower extremity by lifting it off the mat
  4. Flexing one upper extremity while extending contralateral lower extremity and then alternate to opposite extremities.
     Progress to prone position:
  5. Extending one lower extremity
  6. Extending both lower extremity
  Other Names: Core stability exercises
  Arms: McKenzie Extension with External Limb Loading Protocol
Other: McKenzie Extension Exercise Protocol — Static:
  1. Lying Prone
  2. Lying prone in extension
  3. Sustained extension
  4. Posture correction
     Dynamic:
  5. Extension in lying
  6. Extension in lying with clinician overpressure
  7. Extension mobilization
  8. Extension in standing
Other: Moist Heat — Moist Heating for 10 minutes at lumbar spine in prone position using moist heat packs, heated via hydro-collator.

SUMMARY:
Low back pain is one of the most common problem affecting one's daily living activities.

McKenzie Method of Mechanical Diagnostic Therapy (MDT) is an appealing modality of treatment. McKenzie classified the lumbar back pain into three categories i.e. lumbar postural syndrome, lumbar dysfunction syndrome and lumbar derangement syndrome.

Progressive extension bias limb loading exercises at lumbar region emphasizes on lumbar extensor musculature. The purpose of the current study is to determine the effects of extension biased lumbar limb loading exercises along with McKenzie extension protocols in the management of patients with lumbar derangement syndrome, which will also be a cost effective management option. It will also add to the existing pool of knowledge in the fields of conservative low back pain treatment, physical therapy, orthopedic manual therapy and musculoskeletal medicine.

DETAILED DESCRIPTION:
Low back pain is one of the most common problem affecting one's daily living activities.

Back pain results from multifactorial etiology with anatomical, psychological, physiological and social consequences and it is often classified as acute, sub-acute and chronic according to pain duration. Upto 71% of people with acute low back pain in primary care report persistent symptoms and therefore there is requirement for effective treatments in those who have not recovered after acute phase. Therapeutic exercises, manual therapy, functional training, modalities, traction, endurance training of back extensors, Kinesio-taping, trigger point therapy, deep friction massage are some of the procedures being safely and effectively applied by physical therapists to combat back discomfort or disorder.

McKenzie Method of Mechanical Diagnostic Therapy (MDT) approach was developed by Robin McKenzie who was a physical therapist from New Zealand back in 1950s. MDT is an appealing modality of treatment focusing on five areas of benefit-including reliable assessment, early prognosis, self-treatment, better outcomes and prevention of recurrence. The evaluation also determine who will get benefit from treatment and who will require another treatment protocols. McKenzie classified the lumbar back pain into three categories i.e. lumbar postural syndrome, lumbar dysfunction syndrome and lumbar derangement syndrome based on symptomatic or mechanical responses observed during repeated lumbar end range movements. The McKenzie Institute Lumbar Spine Assessment will be used to classify the patients into different syndromes and to choose the desired one fulfilling the inclusion criteria of study.

When normal tissues are deformed over a prolonged period it ends with postural syndrome like slouched posture and the postural syndrome may lead to dysfunction or derangement syndromes. Deformation of structures and tissues that causes pain at end ranges of available motion is characterized as dysfunction syndrome. Derangement syndrome is related to displacement of intervertebral disc with or without involvement of radiating pattern of pain along with back pain and fluctuations in symptoms or pain with directional movements can be observed due to force changes on affected intervertebral disc.

Centralizing and Peripherilizing are two important concepts with a strong association towards derangement syndrome. Centralizing reveals that movements or loading moves the most distal pain proximally while Peripherilizing shows movements or loading moves the pain more distally. McKenzie lumbar extension exercises results in reduction, abolition or centralization of symptoms. In Lumbar derangement syndromes following MDT classification system, a subgroup in which symptoms improve with lumbar extension is labeled as posterior derangement syndrome whereas the subgroup in which symptoms improve with lumbar flexion is labeled as anterior derangement syndrome. Work of many researchers, like Peterson, Machado and Paatelma, provided the strongest evidence regarding the validity of McKenzie method of treatment.

Progressive limb loading exercises at lumbar region fall under two categories, one group emphasis on abdominal musculature and the second group emphasize on lumbar extensor musculature. Patient begins from quadruped position and progress towards prone position initiating with low intensity training and progressing towards greater intensity along with spinal compression in case of lumbar extensors. Progression towards prone position at the end range of motion requires greater control of neutral spine thus providing excellent stabilization of lumbar extensors.

A randomized controlled trial on McKenzie treatment approach in people with chronic low back pain conducted by M.H Halliday et al. provide preliminary evidence that treatment effects of McKenzie Exercises are greater when the core principles are followed with significant reduction in pain and disability of 15.2 [95% CI 7.6 to 22.7] and 11.7 [95% CI 5.4 to18.0]. Srivastav et al. conducted a study at mechanical low back pain with significant improvement having p<0.05 at NPRS & MODI after application of lumbar stabilization exercises along with conventional physical therapy.

An international survey conducted in 15 different countries in 2019 regarding McKenzie classification system involving 64.8% lumbar, 29.6% cervical, 5.6% thoracic spine of 750 patients fulfilling MDT criteria revealed 0.1% postural syndrome, 1.7% dysfunction syndrome, 75.4% derangement and 22.8% other. In derangement syndrome 82.5% were extension biased thus Derangement is the most commonly encountered pain syndrome and extension is so far the most common directional preference.

With the help of this study the investigators can determine the effects of extension biased lumbar limb loading exercises along with McKenzie extension protocols in the management of patients with lumbar derangement syndrome, which will also be a cost effective management option. It will add to the existing pool of knowledge in the fields of conservative spinal management, physical therapy, orthopedic manual therapy and musculoskeletal medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 30 to 50 years
* Patients of both Gender i.e. Male & Female
* Lumbar Derangement Syndrome
* Centralization or Peripheralization phenomenon
* Constant or Intermittent pain worsening on repeated movements
* Somatic, radicular or combination of both patterns of pain
* Positive Radicular signs & symptoms

Exclusion Criteria:

* Lumbar Postural syndrome
* Lumbar Dysfunction syndrome
* Post laminectomy/discectomy
* Spondylolisthesis
* Osteoporosis/Fractures
* Cauda equine syndrome
* Recent history of spinal trauma or surgery
* Lumbar myelopathy
* Patients with known metabolic diseases
* Participants having less than 20% ODI scoring

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 2 weeks
  Oswestry Disability Index (ODI) assess symptoms and severity of low back pain in terms of disablement and the degree to which back pain impacts functional activities. Questionnaire has been designed to give us information as to how one's back or leg pain is affecting his/her ability to manage in everyday life. It has good person and item reliability with an excellent test retest reliability (ICC= 0.97) and floor effect of 29.9% and ceiling effect of 3.9%.
  ODI will be assessed at the base line and at the end of 2 weeks session. Lower score shows better outcome.
Fall Risk Test | 2 weeks
  Biodex Balance System has a fall risk screening test and conditioning protocol based on well-established science and technology. Screening include analytical balance testing by identifying a potential problem and establishes Z-Score on the basis of mean values.
  Fall risk will be assessed at the base line and at the end of 2 weeks session. Lower score shows better outcome.
Postural Stability Index PSI will be assessed at the base line and at the end of 2 weeks session. | 2 weeks
  Postural stability screening test will be used to determine the postural stability index of the participants.
Range of Motion | 2 weeks
  Lumbar ROM including Forward bending, Backward bending, Right side bending and Left side bending will be measured using Inclinometers.
  ROM will be assessed at the base line and at the end of 2 weeks session. Greater range shows better outcome.
Clinical Test of Sensory Integration of Balance | 2 weeks
  Clinical Test of Sensory Integration of Balance (CTSIB) will be assessed at the base line and at the end of 2 weeks session.
Balance Error Scoring System | 2 weeks
  Balance Error Scoring System (BESS) will be assessed at the base line and at the end of 2 weeks session.
STarT Back Screening Tool | 2 weeks
  The Keele STarT Back Screening Tool (SBST) (9-item version) is a brief validated tool, designed to screen primary care patients with low back pain for prognostic indicators that are relevant to initial decision making.
  STarT will be assessed at the base line and at the end of 2 weeks session.

CONTACTS AND LOCATIONS:
Overall Officials: Shoaib Kayani, DPT, MS-OMPT*, Principal Investigator — Foundation University Islamabad; Muhammad Osama, DPT, MSOMPT, CHPE, ACMEd, PhD*, Study Director — Foundation University Islamabad
Locations (2):
- Pakistan (2):
  - Foundation University Islamabad, Islamabad, Federal
  - Shafi International Hospital, Islamabad, Federal

IPD SHARING:
Plan to Share IPD: No